CLINICAL TRIAL: NCT00858585
Title: Genetic Risk of Osteonecrosis of the Jaw (ONJ) in Patients With Metastatic Cancer: Concordance Study
Status: Completed | Type: Observational
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: UMCC 2008.066; HUM 22831 (Other: IRBMED)
Record Dates: First submitted 2009-03-07; First posted 2009-03-10 (Estimated); Last update posted 2019-10-10 (Actual); Status verified 2019-10

CONDITIONS: Breast Cancer
Keywords: Bone metastasis, SNP concordance
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Retained samples will consist of a portion of the specimens collected for this concordance study: peripheral blood leukocytes, lymph nodes, and tumor tissue. All retained samples will be completely de-identified and re-numbered.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study will examine genes in three different tissues and look for similarities and differences between normal cells and cancer cells. The tissues to be studies come from blood, lymph node and cancer.

DETAILED DESCRIPTION:
Subjects will be given an informed consent to read and sign The medical chart will be reviewed for diagnosis and treatment history Blood (about 4 tablespoons) will be drawn at a clinically available time. The lymph node and breast tumor tissue in the University of Michigan pathology repository will be used for research purposes

ELIGIBILITY:
Inclusion Criteria:

* Age at least 18 years of age
* Able to read and sign the informed consent
* Able to provide specimens: one blood draw for white blood cells, provide permission to use tissue already collected.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: breast cancer patients
Sampling Method: Probability Sample
Enrollment: 149 (Actual)
Dates: Start 2009-03; Primary Completion 2011-05 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Single nucleotide polymorphisms | time-independent
  Determine single nucleotide polymorphism concordances between the three DNA specimen sources

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Van Poznak, MD, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States